CLINICAL TRIAL: NCT03996148
Title: Time to Post-Anesthesia Neurological Evaluation and Hemodynamic Stability in Carotid Endarterectomy Comparing Three General Anesthetic Techniques Targeted to a Preset Bispectral Index Value: a Pilot Study
Brief Title: Time to Post-Anesthesia Neurological Evaluation With Three Different Anesthetic Techniques
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Cooper Health System (Other)
Responsible Party: Principal Investigator, Rhea Temmermand, Principal Investigator, The Cooper Health System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17-108
Record Dates: First submitted 2019-05-29; First posted 2019-06-24 (Actual); Results first posted 2022-04-06 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Carotid Artery Stenosis
MeSH Terms: conditions — Carotid Stenosis | interventions — Remifentanil; Propofol; Desflurane; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Remifentanil, Propofol, and Desflurane (Active Comparator): Study group A: no midazolam given; maintenance drugs started immediately after induction and airway is secured.
  Interventions: Drug: Remifentanil, Propofol, and Desflurane
- Remifentanil, Dexmedetomidine, and Desflurane (Active Comparator): Study group B: no midazolam given; maintenance drugs started immediately after induction and airway is secured.
  Interventions: Drug: Remifentanil, Dexmedetomidine, and Desflurane
- Remifentanil and Desflurane (Active Comparator): Study group C (control group): no midazolam given; maintenance drugs started immediately after induction and airway is secured.
  Interventions: Drug: Remifentanil and Desflurane

INTERVENTIONS:
Drug: Remifentanil, Propofol, and Desflurane — Remifentanil - titratable; initial starting dose 0.05 mcg/kg/min Propofol - titratable; initial starting dose 75 mcg/kg/min Desflurane 0.5 MAC
  Other Names: Ultiva; Diprivan; Suprane
  Arms: Remifentanil, Propofol, and Desflurane
Drug: Remifentanil, Dexmedetomidine, and Desflurane — Remifentanil - titratable; initial starting dose 0.05 mcg/kg/min Dexmedetomidine - titratable; initial starting dose 0.5 mcg/kg/hr Desflurane 0.5 MAC
  Other Names: Ultiva; Suprane; Precedex
  Arms: Remifentanil, Dexmedetomidine, and Desflurane
Drug: Remifentanil and Desflurane — Remifentanil - titratable; initial starting dose 0.05 mcg/kg/min Desflurane - titratable
  Other Names: Ultiva; Suprane
  Arms: Remifentanil and Desflurane

SUMMARY:
The objective of this pilot study is to analyze the differences in time to first postoperative neurological examination (cranial nerve XII - tongue movement, movement of extremities) and intraoperative hemodynamic stability with three different general anesthetic techniques that are used for carotid endarterectomy. Carotid endarterectomy surgery removes the plaque and stenosis but has a 1-3% risk of periprocedural stroke or death. The ability to detect neurological abnormalities early after surgery is vital in this patient population to facilitate timely additional diagnostics or interventions if a potential stroke is detected. Anesthetic techniques that facilitate an earlier reliable neurological exam will thus greatly benefit this surgical patient population. The primary objective of this pilot study is to determine the time difference from end of surgery to first neurologic exam between three commonly used anesthetic methods for carotid endareterectomy.

DETAILED DESCRIPTION:
Carotid endarterectomy reduces the incidence of stroke in people with symptomatic, severe carotid artery stenosis. However, there are risks associated with this procedure such as stroke from carotid clamping with poor collateral brain circulation or embolization of carotid plaque debris (Sheth, 2017). Few surgeons monitor the brain during the procedure using SSEP or EEG, as most rely on intraoperative blood pressure management, shunting, and postoperative neurological exam (De Santis, 2016; Kobayashi, 2011).

A Cochrane review of regional versus general anesthesia for carotid endarterectomy reveals no significant difference in outcomes (Vaniyaping, 2013). It is common practice at Cooper Hospital to deliver general anesthesia. The general anesthetic given may affect the length of time to first post-operative neurological response and the hemodynamic stability, though this is not well studied.

A search in PubMed in April 2017 for "carotid endarterectomy AND (general anesthesia OR total intravenous anesthesia OR regional anesthesia) AND neurologic exam" ("endarterectomy, carotid"[MeSH Terms] OR ("endarterectomy"[All Fields] AND "carotid"[All Fields]) OR "carotid endarterectomy"[All Fields] OR ("carotid"[All Fields] AND "endarterectomy"[All Fields])) AND (("general anaesthesia"[All Fields] OR "anesthesia, general"[MeSH Terms] OR ("anesthesia"[All Fields] AND "general"[All Fields]) OR "general anesthesia"[All Fields] OR ("general"[All Fields] AND "anesthesia"[All Fields])) OR (total[All Fields] AND ("intravenous anaesthesia"[All Fields] OR "anesthesia, intravenous"[MeSH Terms] OR ("anesthesia"[All Fields] AND "intravenous"[All Fields]) OR "intravenous anesthesia"[All Fields] OR ("intravenous"[All Fields] AND "anesthesia"[All Fields]))) OR ("regional anaesthesia"[All Fields] OR "anesthesia, conduction"[MeSH Terms] OR ("anesthesia"[All Fields] AND "conduction"[All Fields]) OR "conduction anesthesia"[All Fields] OR ("regional"[All Fields] AND "anesthesia"[All Fields]) OR "regional anesthesia"[All Fields])) AND (neurologic[All Fields] AND exam[All Fields]) revealed no studies comparing anesthetic types and time to first post-operative neurological response in this surgical population. Through anecdotal experience at Cooper Hospital, patients are noted to emerge faster and follow commands sooner when not given preoperative midazolam and given a combined Total Intravenous Anesthetic (TIVA) and volatile inhalational anesthetic technique titrated to a bispectral index (BIS) of 50-60.

Ruling out anesthetic causes of abnormal neurological function is vital in this patient population. Neurological dysfunction that is surgical in nature may require early intervention such as surgical reexploration or CT scan. "Time is brain", and a few minutes difference is enough to cause permanent neurological damage if a progressing stroke is not quickly identified. Anesthetic techniques that demonstrate a quicker return to baseline neurological function will greatly benefit this surgical patient population.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age and older
2. Having carotid endarterectomy surgery
3. Able to undergo a preoperative neurological exam

Exclusion Criteria:

1. Pregnant patients
2. Prisoners
3. Patients with dementia or reduced mental status acute or chronic
4. Known brain tumor or head trauma
5. Known severe, uncorrected coronary artery disease (CAD)
6. Ejection fraction (EF) less than 15%
7. Patients with intraaortic ballon pump (IABP) or other mechanical circulatory assist device
8. Patients with severe chronic obstructive pulmonary disease (COPD)
9. Combined surgical procedures (CABG and CAD)
10. Patients with uncontrolled or severe anxiety requiring benzodiazepine administration
11. Patients with history of difficult airway
12. Sedation other than propofol, dexmedetomidine or volatile anesthetic agent (VAA) is needed for patient (i.e. ketamine in patients with history of neuropathic pain)
13. Intubated or unconscious patients
14. Patients on methadone or fentanyl patch
15. Patients with known unusual or extreme anesthetic requirements
16. Patients who would require an unusual amount of narcotic to control pain
17. Patients having endarterectomy wherein surgeon requests local-regional anesthesia only
18. Patients with known history of prolonged emergence from anesthesia
19. Morbidly obese patients (BMI >40)
20. Patients with scalp or forehead defects that prohibit application of BIS monitor strip

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-09-29 (Actual); Primary Completion 2018-09-19 (Actual); Study Completion 2018-09-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rhea Temmermand, CRNA, Study Director — Cooper University Healthcare
Locations (1):
- Cooper University Hospital, Camden, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Remifentanil, Propofol, and Desflurane | Remifentanil, Dexmedetomidine, and Desflurane | Remifentanil and Desflurane
Started | 7 | 7 | 7
Completed | 7 | 6 | 7
Not Completed | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Remifentanil, Propofol, and Desflurane | Remifentanil, Dexmedetomidine, and Desflurane | Remifentanil and Desflurane | Total
Number analyzed (Participants) | 7 | 6 | 7 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 70 (4) | 73 (12) | 70 (10) | 71 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 1 | 4
  Male | 6 | 4 | 6 | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 7 | 6 | 7 | 20
Preoperative Short Blessed Test [Median (Inter-Quartile Range); unit: units on a scale] — The Short Blessed Test (SBT) is used as a screening test for cognitive changes. There is no unabbreviated scale name. The SBT is a sum of wrong answers (errors) on 6 verbal questions, where each of these is multiplied by a weighting factor. The total score is a whole number ranging from 0 to 28. Based on clinical research findings, the following cut points have been described: 0-4: normal cognition; 5-9: questionable impairment; 10 or more: impairment consistent with dementia or dementing disorder.
  units on a scale | 4 [2 to 6] | 0 [0 to 4] | 5 [1.5 to 10.5] | 4 [2 to 6]
Confusion Assessment Method (3D CAM) [Count of Participants; unit: Participants] — The 3-Minute Diagnostic Interview for Confusion Assessment Method (3D-CAM) is a brief verbal assessment tool for delirium via a short interview of 22 questions. If any answer to the questions is wrong or an observational item is present, a checkmark is applied against one of 4 features that characterize delirium: 1) acute onset or fluctuating course; 2) inattention; 3) disorganized thinking; and 4) altered level of consciousness. If at least one checkmark is present in both domains 1 and 2, and at least one in EITHER 3 or 4, delirium is present.
  Data is # of subjects WITH baseline delirium.
  Participants | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Time to First Neurological Exam
Description: Time to first neurological exam after emergence from general anesthesia
Time Frame: up to 1 hour after emergence from general anesthesia.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Remifentanil, Propofol, and Desflurane | Remifentanil, Dexmedetomidine, and Desflurane | Remifentanil and Desflurane
Number analyzed (Participants) | 7 | 6 | 7
Minutes | 9 (4) | 7 (4) | 7 (3)

ADVERSE EVENTS:
Time Frame: 30 days after enrollment
Arm/Group | Remifentanil, Propofol, and Desflurane | Remifentanil, Dexmedetomidine, and Desflurane | Remifentanil and Desflurane
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 1/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/7 | 0/7 | 0/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Remifentanil, Propofol, and Desflurane (N=7) | Remifentanil, Dexmedetomidine, and Desflurane (N=7) | Remifentanil and Desflurane (N=7)
SAE (Nervous system disorders) | 0 | 1 | 0 — Not study related, stroke

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-03): https://cdn.clinicaltrials.gov/large-docs/48/NCT03996148/Prot_SAP_002.pdf